CLINICAL TRIAL: NCT01879228
Title: A Randomized, Double-blind, Placebo Controlled Study of the Effectiveness of Chronic Incretin-based Therapy on Insulin Secretion in Cystic Fibrosis
Brief Title: Effect of Chronic Incretin-based Therapy in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Michael R. Rickels, MD, MS, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 818014
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Cystic Fibrosis; Pancreatic Insufficiency
Keywords: Cystic Fibrosis; Diabetes; Pancreatic Insufficiency
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency; Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental): The dose of sitagliptin (Januvia®) 100 mg tablet will be taken orally each morning for 6 months.
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo tablet will be taken orally each morning for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — The GPA test as described in the primary outcome section will be performed at baseline and after 6 months of therapy in the Sitagliptin and placebo arms. Furthermore, evaluation of endogenous GLP-1 levels will be assessed by a mixed meal tolerance test compared at baseline and 6 months.
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — The GPA test as described in the primary outcome section will be performed at baseline and after 6 months of therapy in the Sitagliptin and placebo arms. Furthermore, evaluation of endogenous GLP-1 levels will be assessed by a mixed meal tolerance test compared at baseline and 6 months.
  Arms: Placebo

SUMMARY:
In recent years, diabetes has emerged as one of the most significant co-diseases that many Cystic Fibrosis (CF) patients develop. Type 1 and Type 2 diabetes results when either the body does not make enough insulin or the body does not respond correctly to this insulin. Insulin is a hormone which is made by cells in the pancreas and helps carry glucose (sugar) from the food we eat to the cells of the body for energy. While cystic fibrosis related diabetes (CFRD) has many features similar to both Type 1 and Type 2 diabetes, it is very different; therefore, treatment and care of CFRD is not the same.

The purpose of this research study is to examine and understand the various mechanisms that contribute to CFRD and gain a better understanding of potential means to treat CFRD. The primary objective is to determine effectiveness of chronic incretin-based therapy vs. placebo on insulin secretion in CF patients with indeterminate glucose tolerance, impaired glucose tolerance, or CFRD.

DETAILED DESCRIPTION:
Insufficient incretin action has been associated with T2D. To study the possible link between insufficient incretin action and impaired insulin secretion in CFRD as in T2D, the present study will determine whether early intervention with incretin-based therapy using the DPP-4 inhibitor sitagliptin (Januvia®) to raise endogenous levels of the incretin hormones--i.e.--glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotrophic polypeptide (GIP) for a 6-month period will improve insulin secretion in CF patients with indeterminate glucose tolerance, impaired glucose tolerance or early CFRD.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF, defined by positive sweat test or CFTR mutation analysis according to CFF diagnostic criteria
* Age ≥ 18y on date of consent
* Pancreatic insufficiency
* Recent OGTT consistent with Indeterminate-GT, IGT, CFRD w/o fasting hyperglycemia, or an established diagnosis of CFRD without fasting hyperglycemia
* For female subjects, negative urine pregnancy test at enrollment.

Exclusion Criteria:

* Established diagnosis of non-CF diabetes (i.e. T1D) or CFRD with fasting hyperglycemia, (fasting glucose > 126 mg/dL)
* History of clinically symptomatic pancreatitis within last year,
* Prior lung or liver transplant,
* Severe CF liver disease, as defined by portal hypertension,
* Fundoplication-related dumping syndrome,
* Medical co-morbidities that are not CF-related or are unstable per investigator opinion (i.e. history of bleeding disorders, immunodeficiency),
* Acute illness or changes in therapy (including antibiotics) within 6 weeks prior to enrollment,
* Treatment with oral or intravenous corticosteroids within 6 weeks of enrollment,
* Hemoglobin <10g/dL, within 90 days of Visit 1 or at Screening,
* Abnormal renal function, within 90 days of Visit 1 or at Screening; defined as Creatinine clearance < 50 mL/min (based on the Cockcroft-Gault formula) or potassium > 5.5mEq/L on non-hemolyzed specimen,
* A history of anaphylaxis, angioedema or Stevens-Johnson syndrome,
* Inability to perform study specific procedures (MMTT, GPA),
* Subjects, who in study team opinion, may be non-compliant with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-06; Primary Completion 2019-12 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Rickels, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Children's Hospital of Philadelphia and University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kelly A, Sheikh S, Stefanovski D, Peleckis AJ, Nyirjesy SC, Eiel JN, Sidhaye A, Localio R, Gallop R, De Leon DD, Hadjiliadis D, Rubenstein RC, Rickels MR. Effect of Sitagliptin on Islet Function in Pancreatic Insufficient Cystic Fibrosis With Abnormal Glucose Tolerance. J Clin Endocrinol Metab. 2021 Aug 18;106(9):2617-2634. doi: 10.1210/clinem/dgab365. Epub 2021 May 22. PMID 34406395
- See also: Published paper for this study titled: "Effect of Sitagliptin on Islet Function in Pancreatic Insufficient Cystic Fibrosis With Abnormal Glucose Tolerance". — https://pubmed.ncbi.nlm.nih.gov/34406395/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablet will be taken orally each morning for 6 months.
  Sitagliptin: The GPA test as described in the primary outcome section will be performed at baseline and after 6 months of therapy in the Sitagliptin and placebo arms. Furthermore, evaluation of endogenous GLP-1 levels will be assessed by a mixed meal tolerance test compared at baseline and 6 months.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Second-phase Insulin Response Derived From the Glucose-potentiated Arginine Test as a Measure of β-cell Sensitivity to Glucose at Baseline and at 6 Months
Description: The key endpoint of interest will be the change in second phase insulin response derived from the Glucose-Potentiated Arginine (GPA) test. The GPA test will measure insulin, which will be a measure of pancreatic endocrine function in response to the injection of arginine. Arginine is a naturally occurring amino acid (substance) in the body. It will be given in the veins to make the pancreas secrete insulin. After the first injection of arginine, a glucose infusion will be started in order to raise the level of sugar in the blood to 230 mg/dl. Once the level is achieved, arginine will be injected again and blood samples are measured. After a 2 hour break, the glucose infusion will be started to achieve a blood sugar of 340 mg/dl and the arginine injection will be repeated. Comparison of responses at baseline and after 6 months of incretin-based therapy (Sitagliptin) or placebo will be performed using statistical methods.
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: Insulin230 µU/mL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 12 | 12
Insulin230 µU/mL
  Baseline | 0.11 [0.05 to 0.906] | 0.055 [0.022 to 0.13]
  6 Months | 0.085 [0.024 to 0.459] | 0.053 [0.025 to 0.128]

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/13 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=13) | Placebo (N=13)
Mild allergic reaction to study drug (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash or mild allergic reaction to the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT01879228/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT01879228/ICF_001.pdf